CLINICAL TRIAL: NCT04131335
Title: Patient Satisfaction and Dry Symptoms in NHS Patients Undergoing Routine Uncomplicated Cataract Surgery Treated With Prophylactic Phosphate-free, Preservative-free Lubricant Eye Drops. A Randomised Controlled Prospective Study.
Brief Title: Use of Prophylactic Lubricating Drops After Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: City, University of London (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 265860
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye; Cataract Surgery; Patient Related Outcome Measures; Patient Satisfaction
MeSH Terms: conditions — Dry Eye Syndromes; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Experimental arm receives lubricant eye-drops (phosphate-free, preservative-free lubricant eye drops containing 0.15% Sodium Hyaluronate with vitamins A and E (AEONTM Repair) to be administered four times a day for 6 weeks following cataract surgery (in addition to the usual post-operative topical medications of Chloramphenicol 0.5 % eye drops for 1 week and topical dexamethasone 0.1% eyedrops (Maxidex) four times a day for 4 weeks).
  Interventions: Drug: AEONTM Repair; Other: Routine post-operative eye drops used.
- Control Arm (Active Comparator): The control arm group receive the usual post-operative topical medications of Chloramphenicol 0.5 % eye drops for 1 week and topical dexamethasone 0.1% eyedrops (Maxidex) four times a day for 4 weeks after cataract surgery.
  Interventions: Other: Routine post-operative eye drops used.

INTERVENTIONS:
Drug: AEONTM Repair — Lubricating eye drops
  Arms: Experimental Arm
Other: Routine post-operative eye drops used. — Dexamethasone 0.1% eye drops QDS for 4 weeks Chloramphenicol 0.5% eye drops QDS for 1 week

SUMMARY:
This is a randomised controlled trial to assess the use of prophylactic lubricant eye-drops for 6 weeks following uncomplicated, routine cataract surgery to improve patient satisfaction and symptoms of dry eye, compared to controls.

DETAILED DESCRIPTION:
On entry into the study patients will be randomized to receive either lubricant eye-drops (phosphate-free, preservative-free lubricant eye drops containing 0.15% Sodium Hyaluronate with vitamins A and E (AEONTM Repair) to be administered four times a day for 6 weeks following surgery (in addition to the usual post-operative topical medications of Chloramphenicol 0.5 % eye drops for 1 week and topical dexamethasone 0.1% eyedrops (Maxidex) four times a day for 4 weeks) or no additional lubricant drops in addition to the usual medications described above

ELIGIBILITY:
Inclusion Criteria:

* Bilateral or unilateral cataracts requiring surgical intervention
* Age over 18 years
* Able to understand informed consent and the objectives of the trial
* Not pregnant, not breast feeding
* No previous eye surgery

Exclusion Criteria:

* age-related macula degeneration
* glaucoma
* previous retinal vascular disorders
* previous retinal detachment or tear
* any neuro-ophthalmological condition
* any inherited retinal disorder or pathology
* previous strabismus surgery or record of amblyopia
* previous TIA, CVA or other vaso-occlusive disease
* already enrolled in another study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2019-10-14 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction (CatPROM 5) | 6 weeks
  Validated patient satisfaction questionnaire are used. Specially designed and validated conversion tables are used to convert raw scores from questionnaires to Rasch calibrated measures.
Self-reported Health Outcome | 6 weeks
  A validated self-reported health questionnaire is used where a descriptive and vertical Visual Analogue Scale (VAS) are used. The descriptive scale assesses 5 domains at three levels of difficulty (no / some / extreme problems). The VAS is used to to record patients' self-reported health on a scale from 0-100 (100/100 being excellent health, 0/100 being very poor health.
Patient Reported Symptoms (Speed II questinnaire) | 6 weeks
  A validated questionnaire is used with a grading system to grade severity of dry eye . symptoms. Score out of 28. Higher the score, the more significant the dry eye symptoms.

SECONDARY OUTCOMES:
Visual Acuity | 6 weeks
Cornea and Conjunctival Staining Scores | 6 weeks
  The Oxford Scale is used to grade staining of the conjunctiva and cornea. 0-5 (0 no staining, 5 significant staining).
Schirmer 1 test | 6 weeks
  Evaluation of aqueous tear production. Score of more than 10mm is normal. Less than 10mm indicates aqueous tear deficiency .
Tear Break up Time | 6 weeks
  Score of more than 10 seconds is normal. Less than 10 seconds indicates tear evaporative eye disease
Cataract incision site and size | 6 weeks
  Assess cataract incision size in relation to other tests and symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- St Thomas' Hospital NHS Trust London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No